CLINICAL TRIAL: NCT03288324
Title: A 3-part Open-label Study Assessing Safety, Tolerability, Pharmacokinetic and -Dynamic Profiles, and Efficacy of Tofacitinib in Young Adults From Age 18 to 45 With Moderate to Severe Skin Involvement Due to Lupus
Brief Title: Open-label Study of Tofacitinib for Moderate to Severe Skin Involvement in Young Adults With Lupus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WI211648
Record Dates: First submitted 2017-08-29; First posted 2017-09-20 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cutaneous Lupus; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tofacitinib Arm (Experimental): open-label study
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib 5 mg twice daily
  Other Names: Xeljanz

SUMMARY:
This 76-week, 3-part Phase 1b/2 study is intended to evaluate the pharmacological properties (pharmacokinetics and pharmacodynamics), safety, tolerability and preliminary effectiveness of TOFA administrated to young adults (18-45 years) with moderately to severely active SLE-CL. Subjects will be studied at the Cincinnati Children's Hospital Medical Center (CCHMC) and in Cleveland at MetroHealth Medical Center.

DETAILED DESCRIPTION:
Cohort 1 (n=10, weight > 40kg and age > 18 years and ≤ 45 years ) will undergo intense PK-sampling to determine exposures following TOFA dosed at 5 mg BID. TOFA dose escalation will not be considered for inadequate response of SLE-CL.

Cohort 2 (n=10, weight > 40kg and age > 18 years and ≤ 45 years) will be treated with the same dose as Cohort 1. No PK sampling will occur for Cohort 2. Enrollment of Cohort 2 will only start once Cohort 1 has completed 8 weeks of TOFA and results of PK analyses from Cohort 1 are available.

* Part A (up to week 8) requires stable background medications;
* Part B (up to week 24) allows for tapering of corticosteroids (CS) in the setting of significant clinical improvement of SLE-CL as defined by a decrease in Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) activity score by >50% from baseline , and
* Part C (until week 76) permits tapering of other background medications in subjects with clinical remission of SLE-CL (CLASI activity score=0). TOFA dosing is kept stable during Part C.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 years of age and < 45 years of age and > 40 kg body weight.
2. Fulfilled at least 4 out of the 11 Classification Criteria for SLE by the time of screening.
3. Willing to give written informed consent, must fully understand the requirements of the trial, and must be willing to comply with all trial visits and assessments.
4. CLASI activity score of 8 or higher at screening and baseline despite standard of care therapy.
5. Stable dose of prednisone of ≤ 20 mg/day within 2 weeks of enrollment.
6. Female subjects of childbearing potential must use a highly effective method of contraception to prevent pregnancy (abstinence is considered highly effective) and must agree to continue to practice adequate contraception for the duration of their participation in the trial and for 28 days after their last dose of TOFA.
7. Female subjects of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at Trial Day 1 before dosing.
8. For subjects receiving leflunomide treatment, total daily dose does not exceed 20 mg.
9. A negative QuantiFERON-TB Gold In-Tube test performed within the 3 months prior to screening, or within the screening period prior to baseline. A negative PPD test can be substituted for the QuantiFERON-TB.
10. Subjects either have protective varicella titers or evidence of having been vaccinated against varicella.

Exclusion Criteria:

1. Mild SLE-CL defined as a CLASI activity score of 7 or lower at screening and baseline.
2. Increase in CS dosing within 2 weeks prior to Trial Day 1, or expected to require an increase in CS dosing during the first 4 weeks of the study.
3. Use of i.v. corticosteroids within 4 weeks prior to Trial Day 1.
4. Increase in dosing of methotrexate, leflunomide, within 4 weeks before Trial Day 1 or expected to require an increase during the first 8-weeks of the study.
5. Increase in dosing of hydroxychloroquine, or chloroquine within 4 weeks before Trial Day 1 or expected to require an increase during the first 8-weeks of the study.
6. Rituximab within 1 year of Trial Day 1.
7. Increase in dosing of any medication or herbal treatment considered to have immunosuppressive properties with 4 weeks before Trial Day 1.
8. Prior treatment with or known intolerability of TOFA.
9. Use of cyclophosphamide (i.v. or oral), cyclosporine, or tacrolimus within 12 weeks prior to Trial Day 1.
10. Treatment with other investigational agents within the last 6 months or 5 half-lives, or as per washout requirement from the previous protocol, whichever is longer.
11. Estimated glomerular filtration rate less than or equal to 60 mL/min /1.73 m2.
12. Known positive Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV), or Hepatitis B surface antigen (HBsAg) serology.
13. Any condition, including findings in the laboratory tests, medical history, or other screening assessments, that, in the opinion of the Investigator, constitutes an inappropriate risk or a contraindication for participation in the trial or that could interfere with the trial's objectives, conduct, or evaluation.
14. Active central nervous system SLE deemed to be severe or progressive and/or associated with significant cognitive impairment leading to inability to provide informed consent and/or comply with the protocol.
15. Significant renal disease due to a reason(s) other than Lupus Nephritis (e.g. diabetes mellitus, renovascular disease, or antiphospholipid syndrome).
16. Severely active Lupus Nephritis defined as a renal BILAG A score.
17. History of dialysis within 3 months prior to Trial Day 1 or expected to need during the trial.
18. History of or planned renal or other organ transplantation.
19. Known active clinically significant viral, bacterial or fungal infection, or any major episode of infection requiring hospitalization or treatment with parenteral anti-infectives within 8 weeks of screening, or completion of oral anti-infectives within 2 weeks of Trial Day 1.
20. Breastfeeding or currently pregnant.
21. Legal incapacity or limited legal capacity to provide informed consent or assent.
22. Blood dyscrasias, including:

    * Hgb <10 g/dL or Hct <33%.
    * WBC <3.0 x 109/L.
    * Neutrophil count <1.2 x 109/L.
    * Platelet count <100 x 109/L.
    * Lymphocyte count of <0.5 x 109/L.
23. AST or ALT > 1.5 times the upper limit of normal or any other clinically significant laboratory abnormality.
24. History of any other rheumatic autoimmune disease.
25. Infections:

    * Latent or active TB or any history of previous TB.
    * Chronic infections.
    * Any infection requiring hospitalization, parenteral antimicrobial therapy or judged to be opportunistic by the investigator within the 6 months prior to the first dose of study drug.
    * Any treated infections within 2 weeks.
    * History of recurrent (more than one episode) herpes zoster or disseminated (a single episode) herpes zoster or disseminated (a single episode) herpes simplex.
    * History or current symptoms suggestive of any lymphoproliferative disorder, including Cytomegaly Virus (CMV) or Epstein Barr Virus (EBV) related lymphoproliferative disorder, history of lymphoma, leukemia, or signs and symptoms suggestive of current lymphatic disease.
26. Subjects taking potent and moderate cytochrome P450 3A4 (CYP3A4) inhibitors (see Appendix 2).
27. Subjects taking potent and moderate CYP3A4 inducers (see Appendix 2).
28. Subjects who have been vaccinated with live or attenuated vaccines within the 6 weeks prior to the first dose of study medication. All subjects should be up-to-date with respect to standard of care vaccinations (as defined by their country health ministry) as permitted by past immunosuppressive therapy for SLE.
29. Subjects with a malignancy or with a history of malignancy with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
30. Subjects with a history or current diagnosis of diverticulitis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hermine Brunner, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (2):
- United States (2):
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 & Cohort 2: Tofacitinib: Tofacitinib 5 mg twice daily
Period: Overall Study
Arm/Group | Cohort 1 & Cohort 2
Started | 12
Completed | 11
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 & Cohort 2: Tofacitinib: Tofacitinib 5 mg twice daily
  Comparison was not planned for Cohort 1 vs Cohort 2. Cohort 1 received pk analysis. Since only 1 subject was enrolled in cohort 2 the study team is completing analysis with the cohorts combined except for those indicated cohort 1 only in the protocol
Arm/Group | Cohort 1 & Cohort 2
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 21.04 (5.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Oral Clearance (CL/F) (Cohort 1 Only)
Description: Apparent total clearance of the drug from plasma after oral administration
Time Frame: Day 5
Population: Tofacitinib PK was collected from in total of 8 patients, PK parameters were generated for N=7 patients. The PK data for one patient was not used when generating the PK parameters and descriptive summaries due to a dosing event error.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (L/hr)
Groups:
- Cohort 1: Tofacitinib: Tofacitinib 5 mg twice daily
Arm/Group | Cohort 1
Number analyzed (Participants) | 7
(L/hr) | 28.4 (23.5)

2. Secondary Outcome: Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Activity Score
Description: Proportion of subjects who achieve a skin response per the validated CLASI
  The Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) activity score consists of two scores. The first summarizes the activity of the disease while the second is a measure of the damage done by the disease. The Activity Score range is 0-70 with the maximum score (70) indicating the worst outcome. The Damage Score range is 0-80 with the maximum score (80) indicating the worst outcome.
Time Frame: weeks 4, 8 and 24 compared to baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 & Cohort 2
Number analyzed (Participants) | 11
score on a scale
  Baseline | 16.55 (8.03)
  Week 4 | 10.91 (8.4)
  Week 8 | 8.64 (7.8)
  Week 24 | 8.82 (7.9)

3. Secondary Outcome: AUCt (Cohort 1 Only)
Description: Area under the plasma concentration-time curve linear scale Median Concentration (ng/mL) per nominal time 0-8 hours.
Time Frame: Day 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng.hr/mL)
Arm/Group | Cohort 1
Number analyzed (Participants) | 7
(ng.hr/mL) | 176 (23.5)

4. Secondary Outcome: Cmax (Cohort 1 Only)
Description: Maximum (or peak) plasma concentration of Tofacitinib
Time Frame: Day 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)
Arm/Group | Cohort 1
Number analyzed (Participants) | 7
(ng/mL) | 51.7 (21.6)

5. Secondary Outcome: Tmax (Cohort 1 Only)
Description: Time to reach maximum (peak) plasma concentration following administration of Tofacitinib
Time Frame: Day 5
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Cohort 1
Number analyzed (Participants) | 7
hr | 1 [.5 to 2]

6. Secondary Outcome: Vz/F (Cohort 1 Only)
Description: Apparent volume of distribution during terminal phase after non-intravenous administration
Time Frame: Day 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Cohort 1
Number analyzed (Participants) | 7
L | 85.2 (25.6)

7. Secondary Outcome: Half-life of Tofacitinib (Cohort 1 Only)
Description: half-life of Tofacitinib
Time Frame: Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Cohort 1
Number analyzed (Participants) | 7
hr | 2.1 (0.321)

8. Secondary Outcome: Safety of Tofacitinib: Nature, Severity, and Frequency of Adverse Events (Cohorts 1 and 2)
Description: Rate and severity of adverse events and lab abnormalities
Time Frame: 76 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Steroid Dose Comparison
Description: Assess steroid sparing properties of Tofacitinib by comparing doses to baseline and rate of steroid discontinuation
Time Frame: 76 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in SLE Disease Activity Index (SLEDAI) Score
Description: Measure Tofacitinib impact on disease activity
Time Frame: 76 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in British Isles Lupus Activity Group (BILAG) Score
Description: Measure Tofacitinib impact on disease activity
Time Frame: 76 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in SKINDEX Score
Description: Quality-of-life measure for patients with skin disease
Time Frame: Baseline, week 24 and week 76
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Patients Global Assessment Score
Description: Quality-of-life measure for patients
Time Frame: Baseline, week 24 and week 76
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 76 weeks
Groups:
- Cohort 1 and 2: Tofacitinib: Tofacitinib 5 mg twice daily
Arm/Group | Cohort 1 and 2
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 and 2 (N=11)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 and 2 (N=11)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1)
Chlamydial infection (Infections and infestations) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Onychomycosis (Infections and infestations) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Staphylococcal infection (Infections and infestations) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (4)
Urinary tract infection (Infections and infestations) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (4)
Vomiting (Gastrointestinal disorders) | 2 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT03288324/Prot_SAP_000.pdf